CLINICAL TRIAL: NCT02176304
Title: Does Injection Site Matter? A Randomized Controlled Trial to Evaluate Efficacy of Knee Intraarticular Injections on Improval of Patient Reported Outcomes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Ariel D. Davila Parrilla, MD, Orthopedic Surgeon, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Knee Injections
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
Keywords: knee; arthritis; injections; corticosteroids
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suprapatellar Knee Injection Site (Active Comparator): Patients will be injected specified dose of lidocaine and depomedrol through suprapatellar-lateral knee entry site.
  Interventions: Drug: Depomedrol; Drug: Lidocaine
- Anterolateral knee injection (Active Comparator): Patients will be injected specified dose of lidocaine and depomedrol through anterolateral knee entry site.
  Interventions: Drug: Depomedrol; Drug: Lidocaine

INTERVENTIONS:
Drug: Depomedrol — Depomedrol 40 mg/ml, 1 ml injected to knee on day one of intervention.
  Other Names: Depomedrol 40 mg/ml
Drug: Lidocaine — Lidocaine 2% soln, 4 ml injected to knee on day 1 of intervention
  Other Names: Lidocaine 2%

SUMMARY:
Knee osteoarthritis is one of the most prevalent orthopedic conditions worldwide. With the aging population, a 40% patient increase is expected to present at clinics with complaints of primary osteoarthritis by 2025. Multiple studies have attempted to establish non-surgical criteria for knee arthritis and usage of resources to avoid major surgery. It has long been accepted as a treatment option for patients who have failed to respond to NSAIDs and other non-surgical therapies to receive intra-articular injections of steroid and anesthesia mixtures to hold off disease progression.

Various studies have compared different sites of injection and the accuracy rate of the injection being within the joint. Recent studies report a 66% accuracy on palpation-guided injection on the anterolateral knee, 93% accuracy on palpation-guided injection on the superolateral portal of the knee, and new studies show an improvement of up to 98% with use of ultrasound guiding software. However, in a health care system with limited resources, providing patients with US-guided injections represented an increased cost of $178.35 per patient as per 2010 Medicare reports.

Therefore, assuming these accuracy rates, we will compare the anterolateral and superolateral portals for knee injection and their clinical effect to monitor if in fact there is a difference in patient reported outcomes. As a secondary analysis, if no difference is found, a strong case for palpation-guided injections versus ultrasound-guided injections can be made.

In this study we will prospectively enroll 60 patients to be divided into two 30 patient groups with primary knee osteoarthritis. Patients that qualify as subjects will be treated with an intraarticular knee injection through an anterolateral portal or a suprapatellar portal as per group in which they are placed. Scores will be given for pain of the injection and of the baseline illness and compared on a subsequent visit to assess self-reported functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include Early osteoarthritis as per Brandt grades, persistent joint pain warranting a clinic visit, no previous injections given, significant pain in visual analog scale, failure of exercise and oral analgesics.

Exclusion Criteria:

* Exclusion criteria include advanced knee osteoarthritis, patients with bloody effusions, the use of warfarin or antiplatelet therapy, presence of any infection, patients with arthritis other than primary osteoarthritis, patients younger than age 25 due to low likelihood of primary arthritis, pregnant females, diabetics with poor glucose control, and patients that have previously been injected in knee(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Short Term Pain improvement | 1 week
Medium Term Pain Improvement | 1 month
Self Reported Patient Scores Improvement | 1 month
  WOMAC and Visual Analog Scale will be used to monitor improvement

SECONDARY OUTCOMES:
Pain on injection site | baseline
  Will compare pain on site of injection on study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel D Davila-Parrilla, MD, Principal Investigator — University of Puerto Rico Orthopedics Department; Antonio Otero-Lopez, MD, Study Director — University of Puerto Rico Orthopedics Department
Locations (1):
- University of Puerto Rico School Of Medicine Outpatient Clinics, San Juan, Puerto Rico